CLINICAL TRIAL: NCT03320603
Title: Administration of PCC in Patients Admitted in Emergency Care Units for Severe Bleeding While Receiving Oral Anticoagulants: Impact of an Expert ECRF on Adherence to Rules of Proper Use and Outcome
Brief Title: Use of Prothrombin Complex Concentrate in Patients Admitted in Emergency Care Units for Severe Bleeding While Receiving Oral Anticoagulants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: OPTIPLEX 2
Record Dates: First submitted 2017-10-10; First posted 2017-10-25 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Emergency Care for Severe Bleeding While on Anticoagulants
MeSH Terms: interventions — Factor IX

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Other): Prospective collection of data on a standard eCRF (without reminders of recommendations). Prothrombin Complex Concentrate given as standard of care.
  Interventions: Other: Prothrombin Complex Concentrate
- Phase 2 (Other): Prospective collection of data on expert data collection tool (expert eCRF reminding recommendations at each step of the management of severe bleeding). Prothrombin Complex Concentrate given as standard of care.
  Interventions: Other: Expert eCRF; Other: Prothrombin Complex Concentrate

INTERVENTIONS:
Other: Expert eCRF — An expert eCRF will be used to guide physicians during the management of patients treated with Vitamin K Agonist or Direct Oral Anticoagulant admitted in emergency units for severe bleeding.
  Arms: Phase 2
Other: Prothrombin Complex Concentrate — Prothrombin Complex Concentrate given as standard of care

SUMMARY:
The study is assessing the impact of an expert eCRF on the management of severe bleeding in the administration of Prothrombin Complex Concentrate in patients treated with oral anticoagulants and adherence to recommendations or experts' consensus

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Receiving oral anticoagulants (VKA or DOAC)
* With a severe bleeding episode meeting at least one of the following criteria
* External hemorrhage which cannot be controlled by usual means or
* Hemodynamic instability: SBP < 90 mmHg or SBP decrease

  * 40 mmHg from usual SBP or mean BP < 65 mmHg or any sign of shock or
* Patient requiring a hemostatic procedure in emergency:

surgery, interventional radiology, endoscopy or

* Need for transfusion of packed red blood cells or
* Hemorrhage jeopardizing the vital or functional prognosis:

  e.g. intracranial hemorrhage, intraspinal hemorrhage, intraocular or retro-ocular hemorrhage, hemothorax, hemoperitoneum, retroperitoneal hemorrhage, hemopericardium, deep muscle hematoma or compartment syndrome, acute digestive hemorrhage, hemarthrosis.
* Admitted in the participating emergency service
* Accepting the collection of his/her own health-related data

Exclusion Criteria:

* Patient participating in another interventional study
* Pregnant or nursing woman
* Patient under supervision or legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Proper Use of PCC Proportion | 20 months
  Proportion of patients for whom the rules of proper use of PCC have been respected

SECONDARY OUTCOMES:
Time to Death | 20 months
  Time to death
Survival Rate | 20 months
  Survival rate
Proportion of Patients with Poor Outcome | 20 months
  Proportion of patients with poor outcome: comparison of phase 1 and phase 2
Predictors of Poor Outcome | 20 months
  Predictors or poor outcome. Potential predictors of poor outcome will be the time from first symptom to admission, the time from first symptom to Prothrombin Complex Concentrate administration, adherence to recommendations regarding proper use of Prothrombin Complex Concentrate, concomitant antiplatelets treatment, medical history or concomitant diseases (cardiac failure, coronary disease, renal failure, diabetes, severe COPD, cancer). For intracranial hemorrhages predictors will include the volume of intracranial hematoma.
Proportion of Patients with Seroconversion | 20 months
  Proportion of Patients with Seroconversion

CONTACTS AND LOCATIONS:
Locations (26):
- France (26):
  - Centre Hospitalier d'Avignon, Avignon
  - Centre Hospitalier Régional Universitaire de Besançon Hôpital Jean Minjoz, Besançon
  - Clinique Médipole Saint-Roch, Cabestany
  - Centre Hospitalier Universitaire de Caen Hôpital Côte de Nacre Service de Réanimation, Caen
  - Centre Hospitalier Universitaire de Caen Hôpital Côte de Nacre Service des Urgences, Caen
  - Centre Hospitalier Chalon-sur-Saône William Morey, Chalon-sur-Saône
  - Hôpitaux Civils de Colmar, Colmar
  - Hospices Civils de Lyon Hopital Edouard Herriot Service des Urgences, Lyon
  - Clinique du Tonkin, Lyon
  - Hospices Civils de Lyon Centre Hospitalier Lyon-Sud Service de Réanimation, Lyon
  - Hospices Civils de Lyon Centre Hospitalier Lyon-Sud Service des Urgences, Lyon
  - Centre Hospitalier Régional Metz-Thionville Hôpital Mercy, Metz
  - Centre Hospitalier Universitaire de Nantes Hôtel-Dieu, Nantes
  - Centre Hospitalier de Pau, Pau
  - Centre Hospitalier de Perpignan, Perpignan
  - Centre Hospitalier Universitaire de Reims Hôpital Maison Blanche, Reims
  - Centre Hospitalier Universitaire de Rennes Hôpital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Rouen Hôpital Charles-Nicolle, Rouen
  - Centre Hospitalier Universitaire de Strasbourg Nouvel Hôpital Civil Service des Urgences, Strasbourg
  - Centre Hospitalier Universitaire de Strasbourg Hôpital de Hautepierre Service de Réanimation, Strasbourg
  - Centre Hospitalier Universitaire de Strasbourg Hôpital de Hautepierre Service des Urgences, Strasbourg
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon
  - Centre Hospitalier Universitaire de Toulouse Hôpitaux Purpan et Rangueil, Toulouse
  - Centre Hospitalier Régional Universitaire de Tours Hôpital Trousseau, Tours
  - Centre Hospitalier de Valence, Valence
  - Groupe Hospitalier de la Haute-Saône Site de Vesoul, Vesoul